CLINICAL TRIAL: NCT06804642
Title: Rehabilitation of Locomotor Function in Parkinson's Disease by Non-invasive Spinal Cord Stimulation
Brief Title: Spinal Cord Stimulation for Parkinson's Disease Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0700
Record Dates: First submitted 2024-12-18; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; spinal cord; freezing gate; rehabilitation; non-invasive stimulation; neuromodulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-invasive spinal neuromodulation training (Experimental): The overall strategy outlined in this proposal is based on previous data from our own group reporting gait improvement in SCI individuals through activation of spinal locomotor networks located in the lumbosacral region that bear the capability of generating full weight-bearing stepping when epidural stimulation is combined with transcutaneous stimulation of the cervical spinal cord (Angeli & Gerasimenko, 2023). Building on our knowledge from SCI patients, the approach in the present study will be to modulate the ascending proprioceptive fibers important for feedback and posture control and to overcome disruptive signals from descending systems, which presumably occur in PD individuals (Sarica et al., 2023), by taking advantage of the intrinsic abilities of the lumbosacral spinal network to generate stepping. This is a prospective non-blinded non-randomized study. All data will be stored for off-line analysis.
  Interventions: Device: Spinal cord transcutaneous stimulation (scTS)

INTERVENTIONS:
Device: Spinal cord transcutaneous stimulation (scTS) — scTS mapping: Each intervention session will be approximately 2 hours each which includes time to place the scTS stimulating pads and other sensors as needed. Participants will be asked to train 3 days per week during the intervention periods so that they achieve at least 12 sessions. In instances in which availability is limited or they must cancel a session, the intervention period will need to be extended slightly (up to a maximum of four weeks) so that they can achieve at least 12 sessions (1-month intervention period) or 24 sessions (2-month intervention periods) of training. The main study interventions are described below.
  Step-scTS:
  Step-scTS is spinal cord transcutaneous stimulation (scTS) targeted for stepping function. The scTS mapping assessment(s) will assist the study team in determining optimized stimulation parameters for each body and f

SUMMARY:
This study explores the use of multifunctional, non-invasive spinal cord transcutaneous stimulation (scTS) to address axial motor symptoms, particularly gait dysfunction, in Parkinson's disease (PD). These symptoms, resistant to levodopa and inadequately managed by deep brain stimulation (DBS), arise from maladaptive spinal network changes. A non-invasive approach like scTS could overcome limitations associated with invasive spinal cord stimulation (SCS), which requires surgical implantation and lacks adaptability in stimulation site adjustments.

Gait dysfunction in PD stems from disrupted interactions between spinal and supraspinal networks. scTS provides a non-invasive alternative, shown to enhance locomotor functions in conditions such as spinal cord injury, stroke, and cerebral palsy. This study hypothesizes that scTS applied at multiple spinal levels-cervical (C3-C4), thoracic (T11-T12), and lumbar (L1, L2-L3)-can synergistically activate locomotor central pattern generators (CPGs) and improve gait and postural control in PD. Additionally, it is hypothesized that proprioceptive input, combined with scTS, can counteract disruptions in spinal networks and restore voluntary movement.

The primary goal is to evaluate the effects of scTS on stepping performance, postural control, and locomotor recovery in PD. Specific objectives include:

1. Enhancing Locomotor Networks

   * Determine optimal scTS parameters for inducing rhythmic stepping in PD patients.
   * Assess interactions between spinal and supraspinal networks during imagined stepping under scTS in a gravity-neutral setting.
2. Improving Postural Networks

   o Evaluate the effectiveness of scTS in restoring postural control and integrating postural-locomotor functions.
3. Facilitating Neuroplasticity for Movement Recovery o Combine scTS with activity-based recovery training to promote adaptive plasticity in spinal and cortical networks, reducing freezing of gait (FOG).

The research will measure scTS's capacity to generate coordinated stepping and postural movements, integrate proprioceptive feedback, and induce long-term improvements in gait parameters. By targeting spinal locomotor and postural systems, scTS offers a novel, non-invasive approach to addressing gaps in the management of PD gait dysfunction. This work has the potential to significantly enhance the quality of life for individuals with PD, providing a safe, adaptable, and patient-centered therapeutic solution.

DETAILED DESCRIPTION:
Background:

Particular motor symptoms of Parkinson's disease (PD) are currently managed using electrical stimulation of deep structures in the brain. While deep brain stimulation effectively improves tremor, rigidity, bradykinesia, and medication-induced dyskinesias, it does not address axial gait symptoms. Gait symptoms are a late-developing phenomenon in the progression of PD and represent a therapeutic challenge given their poor response to levodopa therapy and deep brain stimulation. This problem, related to spinal maladaptive disorganization as part of pathophysiological changes associated with PD (Tisch et al., 2007), can be approached by electrical spinal cord stimulation (SCS) for alleviation of levodopa-resistant motor symptoms of PD (de Andrade et al., 2016). Thus far, only invasive SCS has been investigated for Parkinsonian gait, with paddle electrodes proving to be the most successful method of stimulation (Milekovic et al., 2023).

While few studies have probed spinal cord stimulation for axial PD symptoms, the optimal location(s) to stimulate the spinal cord are currently unknown (Sarica et al., 2023). Invasive SCS with paddle placement is suboptimal in addressing this gap due to three considerable drawbacks: (i) only one location of the spinal cord can be stimulated with each paddle, (ii) the stimulated location cannot be changed after the SCS paddle is placed, and (iii) paddle SCS placement requires surgery with a laminectomy, which harbors significant risks. To address this gap, a non-invasive stimulation paradigm is needed that permits concomitant stimulation of multiple spinal cord sites to map out the effects on gait during daily life activities and allows altering the stimulation location without the need for surgical intervention.

Previous research suggests that non-invasive multifunctional spinal cord transcutaneous stimulation (scTS) is an effective tool for initiating locomotion in healthy individuals (Gerasimenko et al., 2018) as well as for initiation and rehabilitation of locomotor functions in individuals with motor deficits, including spinal cord injury (SCI) (Gerasimenko et al., 2018; Gerasimenko et al., 2015), stroke (Moon et al., 2024), and cerebral palsy (CP) (Singh et al., 2023).

It is hypothesized that scTS applied to cervical (e.g., C3-C4), thoracic (e.g., T11-T12), and lumbar (e.g., L1, L2-L3) levels, activating locomotor CPGs of upper and lower limbs, as well as postural CPGs, will synergistically facilitate locomotor performance in individuals with PD. Additionally, proprioceptive input is required for gait initiation and locomotion (Zemmar et al., 2024, In Review). Based on these observations, it is hypothesized that concomitant stimulation of (i) multiple motor sites and (ii) proprioceptive feedback tracts activating brain stem nuclei, thalamic nuclei, and the cerebral cortex is required to effectively address gait in individuals with PD.

Therefore, activation of spinal locomotor-related systems in combination with activation of lemniscal and brainstem systems is proposed to promote disruption of anti-kinetic oscillatory synchronization in cortico-basal ganglia circuits, resulting in improved voluntary control of movements in individuals with PD.

Objectives:

The main goal of this project is to determine how multifunctional non-invasive spinal cord stimulation affects stepping performance in individuals with Parkinson's disease (PD). The basic premise is that if the spinal locomotor network is maladaptively affected in PD, then spinal neuromodulation of this network using scTS will be sufficient to correct Parkinsonian gait. One of the most classical features of individuals with PD is the very short and rapid stride length during stepping and the inability to initiate and terminate stepping in a timely manner. The hypothesis is that it will be possible to take advantage of the spinal locomotor-related network to overcome disruptive signals generated in Parkinsonian individuals that disrupt the spinal locomotor network. It is currently unknown whether the spinal locomotor network of individuals with PD has sufficient automaticity potential to generate postural control and rhythmic, coordinated weight-bearing stepping with the aid of multi-site scTS stimulation. It is further hypothesized that the sensory input derived from postural and stepping movements, combined with neuromodulation provided by scTS, can overcome disruptive supraspinal descending signals in individuals with Parkinsonian gait.

The first objective is to determine whether a novel multimodal scTS strategy can transform the spinal locomotor networks of individuals with PD to a functional state enabling rhythmic voluntary movement. Specifically, the goal is to define the specificity of site, frequency, and intensity of scTS required to induce stepping movements and volitionally oscillate leg movements in individuals with PD in a gravity-neutral condition. Interactions between spinal and supraspinal networks in facilitating locomotor movements will be examined when individuals with PD imagine rhythmic stepping movements in the presence of scTS in a gravity-neutral condition.

The second objective is to determine whether a novel multimodal scTS strategy can transform the spinal postural networks of individuals with PD to a functional state enabling postural ability. Specifically, the effectiveness of multimodal scTS to control postural stability will be defined, and the effectiveness of multimodal scTS for the regulation of postural-locomotor integration in individuals with PD will be evaluated.

Lastly, the third objective is to determine whether a novel multimodal scTS strategy, combined with activity-based recovery training, can promote adaptive plasticity of the spinal and cortical locomotor-related networks of individuals with PD to recover voluntary control of movement, particularly by reducing freezing of gait (FOG).

Study Design and Research Procedures:

The overall strategy outlined in this proposal is based on previous data reporting gait improvement in individuals with spinal cord injury (SCI) through activation of spinal locomotor networks located in the lumbosacral region, which are capable of generating full weight-bearing stepping when epidural stimulation is combined with transcutaneous stimulation of the cervical spinal cord (Angeli & Gerasimenko, 2023). Building on knowledge from SCI studies, the approach in this study will be to modulate ascending proprioceptive fibers, important for feedback and posture control, and to overcome disruptive signals from descending systems, which presumably occur in individuals with PD (Sarica et al., 2023). This will be achieved by leveraging the intrinsic abilities of the lumbosacral spinal network to generate stepping. This is a prospective non-blinded, non-randomized study. All data will be stored for offline analysis.

Participants will be identified as individuals with Parkinson's disease and Parkinsonian gait symptoms who consent to participate in the study. Participants will take part in multiple assessment and intervention sessions over a 9-12 month period to track gait and postural improvements over time. Each participant will undergo a detailed medical evaluation prior to baseline assessment. Assessments will last up to 4 hours. Following the completion of baseline assessments, participants will begin the first study intervention period. Post-intervention assessments will be performed approximately 1 week between intervention periods. Each intervention training session will last approximately 2 hours. Participants will train 3 days per week during the intervention periods to achieve at least 12 sessions (1-month intervention period) or 24 sessions (2-month intervention periods). The study timeline, descriptions of assessments, and interventions are outlined below:

Initial Visit:

* Medical Evaluation: Includes a review of medical history, discussion of current medical status, and current medications. A study physician may also complete a physical examination.
* Baseline Assessments: Performed prior to interventions.

Months 1-2:

* Intervention 1: Step-scTS in a gravity-neutral device (GND), 3 sessions per week for 1 month.
* Post-Intervention 1 Assessments: Conducted following the intervention.

Months 2-4:

* Intervention 2: Combination of Step-scTS and locomotor training. Includes 2 sessions per week of Step-scTS with body-weight support treadmill training (BWS) and 1 session per week of Step-scTS with overground locomotor training using an assistive device, for a total of 3 sessions per week over 2 months.
* Post-Intervention 2 Assessments: Conducted following the intervention.

Months 4-6:

* Intervention 3: Step-scTS combined with overground locomotor training using an assistive device, 3 sessions per week for 2 months.
* Post-Intervention 3 Assessments: Conducted following the intervention

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease;
* Adults aged 18 to 80 years;
* Competent to give informed consent for the research protocol;
* Able to understand instructions;
* Able to ambulate 10-meters.

Exclusion Criteria:

* Co-morbidities affecting gait;
* Clinically significant cognitive dysfunction;
* Clinically significant depression or major active psychiatric illness such as schizophrenia, bipolar disorder, or major depressive disorder;
* Terminal illness associated with <12-month survival;
* Have a current diagnosis or condition such as major cardiac insufficiency, determined clinically by the study doctors;
* Current alcohol or substance abuse that is uncontrolled or unmanageable;
* Individuals unable to communicate with the investigator and study staff; and/or
* Individuals with any illness that, in the study doctors' opinion, may preclude them from spinal cord transcutaneous stimulation, activity-based recovery training, or participation in study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-12-11 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
A. Assessment of Multisegmental Motor Responses (MMR) | From date of screening until the date of data is analyzed, up to 48 months.
  Multisegmental motor responses in different leg muscles evoked by non-invasive stimulation of the dorsal lumbosacral spinal cord will be recorded. Such responses are the basic components of the lower-limb muscle responses that are elicited by transcutaneous stimulation of posterior lumbar cord structures. Multi-Segmental Motor Responses will be evoked transcutaneously by using a constant current stimulator (Cosyma, Inc. or Digitimer-Constant Current Stimulator, e.g., DS8R) between the C2 spinous process and the Coccyx. Small cathodes (pre-gelled, soft surface electrodes) will be placed over the skin between the C2 spinous process and Coccyx (midline with a single cathode or left and right of midline with a split cathode) while larger anode(s) will be placed over the anterior spine at different levels, at segments just below the cathode, on the abdomen, or along the pelvis.
Spinal Cord Transcutaneous Stimulation (scTS) Mapping electromyography (EMG) | From date of screening until the date of data is analyzed, up to 48 months.
  Mapping will be carried out through assessment of electrophysiological and functional changes. EMG will be used to assess muscle activity. The mapping assessment may take place with the participant in supine, side-lying in a gravity-neutral device, upright while standing, or upright while stepping. Assistance will be provided as needed. A safety limit of 250 mA will be implemented. Other stimulation parameters include: 5-10 kHz carrier frequency for modulation of discomfort from stimulation, 0.25-3.0 ms pulse width duration, and 10-100 Hz.
Spinal Cord Transcutaneous Stimulation (scTS) Mapping electroencephalography (EEG) | From date of screening until the date of data is analyzed, up to 48 months.
  Mapping will be carried out through assessment of electrophysiological and functional changes. EEG will be used to assess brain activity. The mapping assessment may take place with the participant in supine, side-lying in a gravity-neutral device, upright while standing, or upright while stepping. Assistance will be provided as needed. A safety limit of 250 mA will be implemented. Other stimulation parameters include: 5-10 kHz carrier frequency for modulation of discomfort from stimulation, 0.25-3.0 ms pulse width duration, and 10-100 Hz.
Stepping Performance in a Gravity-Neutral Device (GND) with electromyography (EMG). | From date of screening until the date of data is analyzed, up to 48 months.
  Limb coordination and muscle activation during visual imaginary stepping and gravity-neutral ambulation will be assessed with surface EMG of multiple trunk and lower extremity muscles including pelvic stabilizers (quadratus lumborum), hip extensors (gluteus), hip flexors (iliopsoas), knee extensor (rectus femoris), knee flexor (biceps femoris), ankle dorsiflexor (tibialis anterior), and ankle plantar flexor (medial gastrocnemius and soleus) without and with scTS.
Stepping Performance in a Gravity-Neutral Device (GND) with kinematics. | From date of screening until the date of data is analyzed, up to 48 months.
  Limb coordination during visual imaginary stepping and gravity-neutral ambulation will be assessed with gait kinematics determined with goniometers at the top arm, hip, knee, and/or ankle and/or with 3D motion capture.
Stepping Performance in a Gravity-Neutral Device (GND) with plantar stimulation. | From date of screening until the date of data is analyzed, up to 48 months.
  Limb coordination during visual imaginary stepping and gravity-neutral ambulation will be assessed with plantar pressure stimulation (Korvit) to be used based on participant presentation. When used, pressure sensing insoles (Noraxon Ultium) will be placed in orthotics to track inflation under the heel and forefoot and synchronize with other data types.
Stepping Performance in a Gravity-Neutral Device (GND) with electroencephalography (EEG). | From date of screening until the date of data is analyzed, up to 48 months.
  EEG will be recorded before, during, and after scTS. Cortical activity will be correlated with gait performance/limb kinematics.
D. Assessment of Balance and Gait: Tinetti Balance & Gait Test, Rating Instrument to Assess Festination and Freezing Gait, and Push & Release Test | From date of screening until the date of data is analyzed, up to 48 months.
  The Tinetti Balance and Gait Test, also known as the performance-oriented mobility assessment, uses a standardized scoring system to assess participants' balance and gait. The examiner will be near the participant during each part of the assessment in case the participant exhibits any risk of falling. Scoring is ordinal with a range from 0 to 2; 0 indicates severe impairment and 2 indicates independence. For the balance assessment, the participant starts in a seated position on a hard, armless, stable chair and is instructed to rise from seated without using their arms or hands. Once standing, the participant is instructed to move their feet as close together as possible. The examiner then presses on the participant's sternum with their palm three times while the participant's eyes are open and three times while the participant's eyes are closed. During the last component of the balance assessment, the participant is asked to make a 360-degree turn and sit back in the chair.
New Freezing of Gait Questionnaire (NFOG-Q) | From date of screening until the date of data is analyzed, up to 48 months.
  The Freezing of Gait Questionnaire is a six-item scale (range 0-24); four items assess FOG severity, and two items assess general gait difficulties. The New Freezing of Gait Questionnaire was developed to address limitations of the original questionnaire. The NFOG-Q adds an initial item to the original questionnaire; based on the answer to this initial item, part II includes questions about FOG severity, and part III includes questions about impact. The NFOG-Q was found to be test-retest reliability and high agreement between patients with Parkinson's disease and their carers.

SECONDARY OUTCOMES:
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | From date of screening until the date of data is analyzed, up to 48 months.
  The Movement Disorder Society (MDS)-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Task Force revised and expanded the UPDRS. It has four parts: I: Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications. Twenty questions are completed by the participant. The Non-motor Experiences of Daily Living (part I) include questions on cognitive impairment, hallucinations and psychosis, depressed mood, anxious mood, apathy, dopamine dysregulation syndrome, sleep, pain and other sensations, urinary problems, constipation problems, orthostatic hypotension, and fatigue. Motor Experiences of Daily Living (part II) include questions related to speech, saliva and drooling, chewing and swallowing, eating tasks, dressing, hygiene, handwriting, participating in hobbies and other activities, turning in bed, tremor, getting out of bed, walking and balance, and freezing.
Time to Navigate (TTN) Test | From date of screening until the date of data is analyzed, up to 48 months.
  The Time to Navigate (TTN) test was developed as a practical and objective clinical measure of FOG severity. The TTN test involves similar situations as those in the Rating Instrument to Assess Festination and Freezing of Gait with single-tasking and dual-tasking. The TTN does not include navigating through a door but instead includes a longer walking pass and navigating around an object and a narrow corridor. Completing both assessments with participants who opt into participating will allow comparison between the two clinical measures and additional information about participants' functional presentation and what kinds of activities elicit FOG.
Modified Ashworth Scale (MAS) and Range of Motion (ROM) Testing | From date of screening until the date of data is analyzed, up to 48 months.
  The modified Ashworth Scale scores muscle spasticity by assessing the resistance observed during passive muscle stretching. A six-category ordinal scale (0 = no increase in muscle tone; 1 = Slight increase in muscle tone with catch and release; 1+ = Slight increase in tone with catch; 2 = Marked increase in muscle tone but affected parts move easily; 3 = considerable increase in muscle tone and passive movement is difficult; 4 = affected part(s) rigid in flexion or extension) is used to score the participant's spasticity in the muscles of interest. During the MAS, range of motion (ROM) testing will also be completed to track any musculoskeletal abnormalities and/or improvements in ROM. sEMG, fine wire EMG, joint kinematics, and body weight force will be measured.
10-Meter Walk Test | From date of screening until the date of data is analyzed, up to 48 months.
  The 10-meter walk test (10MWT) assesses walking speed in meters per second over a short duration. Assistive devices can be used during this test. Participants will be given space to accelerate to their preferred walking speed before the start of the 10-meter distance. sEMG, fine wire EMG, joint kinematics, and body weight force will be measured. Following an initial 10MWT without stimulation and adequate rest, participants who are able will repeat the test with multi-site scTS.
6-Minute Walk Test | From date of screening until the date of data is analyzed, up to 48 months.
  The 6-minute walk test (6MWT) assesses walking endurance over a specific time window. Assistive devices can be used during this test. Participants will be permitted to take standing breaks during the 6-minute period, but if participants require a seated rest break, the 6MWT will be completed at that point. sEMG, fine wire EMG, joint kinematics, and body weight force will be measured. Following an initial 6MWT without stimulation and adequate rest, participants who are able will repeat the test with multi-site scTS.

OTHER OUTCOMES:
Propriospinal Pathway Assessment (PSPA) | From date of screening until the date of data is analyzed, up to 48 months.
  Propriospinal pathways will be assessed by electrically or magnetically stimulating a variety of peripheral nerves such as, but not limited to, the ulnar, superficial radial, common and superficial peroneal, and femoral nerves. We will then record interlimb reflexes/responses from various muscles at rest. Surface or fine-wire electrodes to record this activity will be utilized. Additionally, nerve stimulation could be paired with various other types of stimulation, which could be the Hoffman reflex, multisegmental motor responses (MMRs), or in the presence of transcutaneous electrical stimulation. Conditioning of these responses will allow us to identify the effects of propriospinal pathways in the human spinal cord under conditions when we typically might not be able to see these responses in resting muscles.
Supraspinal Connectivity Assessment (SSCA) | From date of screening until the date of data is analyzed, up to 48 months.
  Test responses will be evoked using sub maximal transcutaneous electrical spinal cord stimulation of 1 ms duration at intensities of up to 100 mA delivered over the intra-spinous space between the spinous processes of the T10 and Coccyx vertebrae, with participants lying in a supine position. Stimulation will be delivered using Digitimer constant current stimulator (Digitimer Ltd., UK). Reponses will be recorded via surface EMG electrodes placed bilaterally over the proximal and distal lower extremities' muscles. The conditioning stimulation will precede the test pulse to assess the Long propriospinal pathways: Electrical stimulus over the lateral epicondyle as well as between the intra-spinous space between C3 and C5 or ulnar nerve stimulation using a Digitimer constant current stimulator (Digitimer Ltd., UK). The intervals between the conditioning and test stimuli will vary from 5 to 200 ms.
Reticulospinal Pathway Assessment (RSPA) | From date of screening until the date of data is analyzed, up to 48 months.
  The reticulospinal pathway has been attributed to widespread muscle contractions in response to sudden unexpected auditory stimuli. The latency, habituation after repeated stimuli and characteristics of muscular contraction suggest that the most likely mediating structure is the reticular formation in the medulla and pons. Implementing an acoustic startle reaction has been shown to result in muscles responses in facial, arm and sometimes leg muscles that are attributed to the reticulospinal pathways. After SCI it appears that the reticulospinal pathway is strengthened as a compensatory mechanism. The reticulospinal pathway will be evaluated either while the participant is at rest or through paired conditioning studies.
Voluntary Motor Control of Hip, Knee, Ankle, and Toe Assessment | From date of screening until the date of data is analyzed, up to 48 months.
  This novel assessment paradigm was developed to evaluate the state of the corticospinal pathway by using stimulation pulses timed with a task-driven movement attempt. Force levels will be assessed with a force transducer secured to a cable and/or a dynamometer that is attached to the appropriate limb segment and the associated muscle activity patterns will be assessed from surface EMG recordings of the appropriate muscles: hip extensor (gluteus), hip flexor (iliopsoas), knee extensor (rectus femoris), knee flexor (biceps femoris), ankle dorsiflexor (tibialis anterior), and ankle plantar flexors (medial gastrocnemius and soleus). Participants will be lying supine on a bed, supine or seated on an adjustable reclining chair with their leg strapped to a dynamometer to measure force, or side-lying in the GND. Spinal stimulation will be provided over the thoracolumbosacral spinal cord (e.g., between L1-L2 vertebral bodies).
Corticospinal Pathway Assessment (CSPA) with Transcranial Magnetic Stimulation (TMS) | From date of screening until the date of data is analyzed, up to 48 months.
  Transcranial magnetic stimulation (TMS) of the cortex has been used extensively in human to assess the integrity of the descending corticospinal tract. TMS of the cortex has been shown to have prognostic value after human spinal cord injury relating to recovery of function. The corticospinal tract function will be tested by recording motor evoked potentials (MEPs) in various muscles of interest. Single pulse transcranial magnetic stimulation will be administrated using a Magstim. We will use a variety of different coils depending on which muscles we are trying to activate (circular coil, figure-8 coil or double cone coil).
Spinal Magnetic Stimulation Assessment (SMSA) | From date of screening until the date of data is analyzed, up to 48 months.
  Spinal magnetic stimulation is to activate spinal neurons in a painless non-invasive fashion using magnetic stimulation. A figure of 8 or circular coil is placed over a focused segment of the spine between C2 to L4 and a single or a high frequency repetitive magnetic pulse is applied. Motor evoked potentials, EMG and H-reflex responses will be measured. The purpose is to assess the ability of magnetic stimulation to activate spinal neuronal modulation locomotor networks and spinal central pattern generators-measured using EMG. The goal is to optimize parameters for consistent activation of spinal circuitry in a painless non-invasive manner.
Vestibulospinal Pathway Assessment (VPA) | From date of screening until the date of data is analyzed, up to 48 months.
  Galvanic stimulation has been a successful tool to probe vestibular function and the balance system in humans by delivering a perturbation at the receptor level during sitting, standing, walking and running. This non-invasive technique activates the vestibular cortices and adjacent cortical areas by application of weak direct currents, delivered by two electrodes attached to the mastoids. Muscle responses (EMG) are seen only in muscles engaged in balance indicating a task-dependent gating of descending vestibulospinal influences. Bipolar galvanic stimulation (2-4 mA) will be applied over the mastoid processes.
Cutaneomuscular Reflex (CMR) | From date of screening until the date of data is analyzed, up to 48 months.
  Long-lasting cutaneomuscular reflexes can readily be elicited following spinal cord injury by electrically stimulating cutaneomuscular afferents supplying the side and sole of the foot with long pulse trains (300 Hz, 14 pulses, 0.5-ms pulse width. This reflex comprises three components: an early-latency short-lasting polysynaptic reflex component (SPR: onset 50-70 ms after stimulation, and lasting 50 ms); a polyphasic longer-lasting polysynaptic reflex (LPR: end of SPR until 300 ms after stimulation in incomplete SCI participants, start of reflex until 300ms after stimulation in complete SCI participants that do not exhibit SPR) and a later long-lasting reflex component (LLR: 500 ms after stimulation until the end of the reflex response.
Hoffman Reflex (H-reflex) | From date of screening until the date of data is analyzed, up to 48 months.
  The Hoffman reflex (H-reflex), the electrical analogue of the stretch reflex is considered a measure of segmental motor excitability. The modulation of this reflex has been well documented in humans during voluntary contractions of the upper and lower limbs demonstrating the role of supraspinal influence on segmental reflexes. Abnormal modulation of the H-reflex has been shown in humans after neurologic disorders including spastic paraparesis, stroke and spinal cord injury with pre-synaptic inhibition as a prominent mechanism. The H reflex is evoked by electrically or magnetically stimulating a peripheral nerve in your body. This evokes a response in the muscles that are innervated by this nerve. The H-reflex will be used to assess spinal cord excitability in individuals.
Respiratory Motor Control Assessment (RMCA): electromyography (EMG) | From date of screening until the date of data is analyzed, up to 48 months.
  The RMCA will utilize a multi-muscle EMG-based measure of motor output from the central nervous system recorded during voluntary tasks attempted in the sitting position. Participants will be provided with sufficient rest time between maneuvers, and each will be repeated with the goal of obtaining three attempts that can be analyzed. When participants show signs of fatigue or cannot perform a given maneuver, portions of the RMCA will be skipped to ensure their comfort and safety.
Respiratory Motor Control Assessment (RMCA): pulmonary function test (PFT) | From date of screening until the date of data is analyzed, up to 48 months.
  The RMCA will utilize measure of standard PFT attempted in the sitting position. Participants will be instructed on how to perform maneuvers by a trained examiner. Participants will be provided with sufficient rest time between maneuvers, and each will be repeated with the goal of obtaining three attempts that can be analyzed. When participants show signs of fatigue or cannot perform a given maneuver, portions of the RMCA will be skipped to ensure their comfort and safety.
Orthostatic Tilt Table Test: blood pressure changes | From date of screening until the date of data is analyzed, up to 48 months.
  The orthostatic stress test measuring changes in beat-to-beat arterial blood pressure to diagnose orthostatic hypotension. Each participant will be assessed in the morning in a quiet, temperature-controlled (~72oF/22oC) laboratory. Their diet will be restricted to exclude caffeine, alcohol, and foods that are high in fat the evening prior and the morning before the study. Participants will be asked to use the restroom to void their bladder before the assessment begins. Participants will be placed in a cardiac chair (Chair Hydraulics, Steris Corp., Mentor, OH) or on a tilt-table (Hausmann Wheelchair Accessible Hi-Lo Tilt-Table, Patterson Medical, IL). Before the recording begins, each participant will be acquainted with the equipment and study setup.
Orthostatic Tilt Table Test: baroreflex responsiveness changes | From date of screening until the date of data is analyzed, up to 48 months.
  The orthostatic stress test will be utilized to evaluate baroreflex responses by assessing heart rate variability. Each participant will be assessed in the morning in a quiet, temperature-controlled (~72oF/22oC) laboratory. Their diet will be restricted to exclude caffeine, alcohol, and foods that are high in fat the evening prior and the morning before the study. Participants will be asked to use the restroom to void their bladder before the assessment begins. Participants will be placed in a cardiac chair (Chair Hydraulics, Steris Corp., Mentor, OH) or on a tilt-table (Hausmann Wheelchair Accessible Hi-Lo Tilt-Table, Patterson Medical, IL). Before the recording begins, each participant will be acquainted with the equipment and study setup.
Cognitive Assessment Battery (CAB) | From date of screening until the date of data is analyzed, up to 48 months.
  The cognitive assessment battery will be used to measure changes in cognitive capacity by using standard questionnairy.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, MD, Ph.D., Study Director — University of Louisville
Locations (1):
- Frazier Rehab Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no data-sharing plan required for this PI-initiated study.